CLINICAL TRIAL: NCT02805049
Title: Pharmacokinetic Study on Echinocandins for Patients With Septic Shock Following Secondary Peritonitis
Brief Title: Pharmacokinetic Study on Echinocandins for Patients With Septic Shock Following Secondary Peritonitis (EPI Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2016/CR-01; 2016-002708-17 (EudraCT Number)
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2019-01

CONDITIONS: Septic Shock; Peritonitis
MeSH Terms: conditions — Shock, Septic; Peritonitis | interventions — Echinocandins; Caspofungin; Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study population (Experimental): The study population consisted of patients admitted to the ICU for septic shock associated with secondary peritonitis and requiring antifungal therapy via echinocandins (micafungin or caspofungin).
  Interventions: Drug: Echinocandins

INTERVENTIONS:
Drug: Echinocandins — The patients included in this protocol require routine treatment with caspofungin or micafungin. Though this intervention is under study, it is not modified by this protocol.
  Other Names: caspofungin or micafungin

SUMMARY:
The main objective of this study is to describe the pharmacokinetics of the prescribed echinocandins for septic shock with secondary peritonitis for which intra-abdominal fungal infection is suspected or proven.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* Determine whether the current recommended doses of caspofungin achieve the Pharmacokinetic/Pharmacodynamic (PK/PD) target for this molecule.
* Determine whether the current recommended doses of micafungin achieve the PK / PD target for this molecule
* Describe the peritoneal concentrations of echinocandins in secondary peritonitis complicated with septic shock
* Identify via modeling PK / PD parameters and based on monte Carlo simulations the optimal dosing regimen for caspofungin and micafungin in this population

ELIGIBILITY:
Inclusion Criteria:

* The emergency inclusion procedure was correctly applied according to French law (signature of consent form by a patient-designated trusted person or a family member, or a medical decision to proceed with patient inclusion if the latter two persons are unavailable) ---- OR ---- signature of the consent form by the patient
* The patient must be insured or beneficiary of a health insurance plan
* The patient is 18 years of age or older
* The patient has beed admitted to the ICU for septic shock accompanying secondary peritonitis
* Patient requiring antifungal treatment via echinocandins (caspofungin or micafungin)
* A venous or arterial access for blood sampling is already in place for routine care

Exclusion Criteria:

* The patient is participating in an interventional study that may affect the results of the present study, or has participated in such a study within the past 3 months
* The patient is under judicial protection, or is an adult under guardianship
* The patient is pregnant, parturient or breastfeeding
* Moribund patient
* Known positive serology for human immunodeficiency virus (HIV)
* Known positive serology for hepatitis C
* Known diagnosis for tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-28 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Antifungal treatment plasmatic clearance (L/h) | Day 1
Antifungal treatment plasmatic clearance (L/h) | Days 3-5
The volume of distribution (L) corresponding to plasmatic antifungal treatment concentration | Day 1
The volume of distribution (L) corresponding to plasmatic antifungal treatment concentration | Days 3-5
Intercompartmental transfer constant for a bi-compartmental model for plasmatic antifungal treatment concentration | Day 1
Intercompartmental transfer constant for a bi-compartmental model for plasmatic antifungal treatment concentration | Days 3-5
The area under the curve for plasmatic antifungal treatment concentrations | Day 1
The area under the curve for plasmatic antifungal treatment concentrations | Days 3-5
The maximum concentration for plasmatic antifungal treatment concentrations | Day 1
The maximum concentration for plasmatic antifungal treatment concentrations | Days 3-5
The minimum concentration for plasmatic antifungal treatment concentrations | Day 1
The minimum concentration for plasmatic antifungal treatment concentrations | Days 3-5

SECONDARY OUTCOMES:
The target Pharmacokinetic/Pharmacodynamic ratio for caspofungin | Day 1
  corresponds to: area under the curve / minimum inhibitory concentration >865
The target Pharmacokinetic/Pharmacodynamic ratio for caspofungin | Days 3-5
  corresponds to: area under the curve / minimum inhibitory concentration >865
The target Pharmacokinetic/Pharmacodynamic ratio for micafungin | Day 1
  corresponds to: area under the curve / minimum inhibitory concentration >285 et 3000
The target Pharmacokinetic/Pharmacodynamic ratio for micafungin | Days 3-5
  corresponds to: area under the curve / minimum inhibitory concentration >285 et 3000
The area under the curve for peritoneal antifungal treatment concentrations | Day 1
The area under the curve for peritoneal antifungal treatment concentrations | Days 3-5
The maximum concentration for peritoneal antifungal treatment concentrations | Day 1
The maximum concentration for peritoneal antifungal treatment concentrations | Days 3-5
The minimum concentration for peritoneal antifungal treatment concentrations | Day 1
The minimum concentration for peritoneal antifungal treatment concentrations | Days 3-5
The probability of attaining the targeted Pharmacokinetic/Pharmacodynamic ratio | Day 1
The probability of attaining the targeted Pharmacokinetic/Pharmacodynamic ratio | Days 3-5
The fraction of the probability of attaining the targeted Pharmacokinetic/Pharmacodynamic ratio | Day 1
The fraction of the probability of attaining the targeted Pharmacokinetic/Pharmacodynamic ratio | Days 3-5

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- Royal Brisbane Women's Hospital, Herston, Australia
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Garbez N, Mbatchi L, Wallis SC, Muller L, Lipman J, Roberts JA, Lefrant JY, Roger C. Prospective Cohort Study of Micafungin Population Pharmacokinetic Analysis in Plasma and Peritoneal Fluid in Septic Patients with Intra-abdominal Infections. Antimicrob Agents Chemother. 2021 Jun 17;65(7):e0230720. doi: 10.1128/AAC.02307-20. Epub 2021 Jun 17. PMID 33846133